CLINICAL TRIAL: NCT02612155
Title: A Phase II Multi-site Study of Autologous Cord Blood Cells for Hypoxic (HIE)
Brief Title: A Multi-site Study of Autologous Cord Blood Cells for Hypoxic Ischemic Encephalopathy
Acronym: (HIE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Cotten (Other)
Collaborators: The Robertson Foundation (Other)
Responsible Party: Sponsor-Investigator, Michael Cotten, Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00066647
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Moderate or Severe Hypoxic-ischemic Encephalopathy in Newborns
Keywords: Hypoxic-ischemic encephalopathy; autologous cord blood cells; newborn infants
MeSH Terms: conditions — Lymphoma, Follicular; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention cell recipients (Experimental): Experimental: infusions: infants with moderate to severe hypoxic ischemic encephalopathy, begin cooling, and have autologous nucleated cord blood cells available for infusion will receive up to two infusions. Outcomes will be measured at 22-26 months by neurodevelopment assessment
  Interventions: Biological: Infusion of autologous cord blood
- Placebo recipients (Placebo Comparator): Control: infants with moderate to severe hypoxic ischemic encephalopathy, begin cooling, and have cord blood available for infusion will receive placebo (a mix of autologous cord blood red blood cells and plasma) infusions. Outcomes will be measured at 22-26 months by neurodevelopment assessment
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Infusion of autologous cord blood — Infants who meet study enrollment criteria will receive up to 2 infusions of their own volume reduced cord blood cells. The number of doses will be determined by the amount of available cord blood cells.
  Arms: Intervention cell recipients
Biological: Placebo — Infants who meet study enrollment criteria will receive up to 2 placebo infusions composed of an equivalent volume (volume of product that would have been administered if the infant randomized to the intervention arm) of packed red blood cells (PRBCs) from the red cell compartment of the separated cord blood unit.
  Arms: Placebo recipients

SUMMARY:
This study will test the safety and efficacy of an infusion of a baby's own (autologous) umbilical cord blood as compared with placebo in babies born with history and signs of hypoxic-ischemic brain injury.

DETAILED DESCRIPTION:
The purpose of this phase II study is to assess the safety and efficacy of up to two intravenous infusions of autologous volume and red blood cell reduced nucleated umbilical cord blood cells as compared with placebo in neonates with neonatal encephalopathy undergoing hypothermia treatment. Efficacy will be estimated by one year survival and score on Bayley III scores in all three domains equal to or greater than 85. This will be a randomized, double-blind, placebo controlled multi-site trial of up to 160 infants who qualify for cooling.

ELIGIBILITY:
Inclusion Criteria:

1. NICHD Neonatal Research Network Hypothermia Trial inclusion criteria
2. Mothers must have consented or given verbal assent for cord blood collection at delivery, and cord blood must be available for volume and red blood cell reduction before 45 hours of age
3. The infant must be able to receive at least one dose of autologous cord blood before 48 hours of age
4. All infants must have signs of encephalopathy within 6 hours of age

Exclusion Criteria:

1. Major congenital or chromosomal abnormalities
2. Severe growth restriction (birth weight <1800 g)
3. Opinion by attending neonatologist that the study may interfere with treatment or safety of subject
4. Moribund neonates for whom no further treatment is planned
5. Infants born to mothers are known to be HIV, Hepatitis B, Hepatitis C or who have active syphilis or CMV infection in pregnancy
6. Infants suspected of overwhelming sepsis
7. ECMO initiated or likely in the first 48 hours of life

Ages: 0 Hours to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cotten, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Cotten CM, Murtha AP, Goldberg RN, Grotegut CA, Smith PB, Goldstein RF, Fisher KA, Gustafson KE, Waters-Pick B, Swamy GK, Rattray B, Tan S, Kurtzberg J. Feasibility of autologous cord blood cells for infants with hypoxic-ischemic encephalopathy. J Pediatr. 2014 May;164(5):973-979.e1. doi: 10.1016/j.jpeds.2013.11.036. Epub 2013 Dec 31. PMID 24388332
- [Background] Shankaran S, Laptook AR, Ehrenkranz RA, Tyson JE, McDonald SA, Donovan EF, Fanaroff AA, Poole WK, Wright LL, Higgins RD, Finer NN, Carlo WA, Duara S, Oh W, Cotten CM, Stevenson DK, Stoll BJ, Lemons JA, Guillet R, Jobe AH; National Institute of Child Health and Human Development Neonatal Research Network. Whole-body hypothermia for neonates with hypoxic-ischemic encephalopathy. N Engl J Med. 2005 Oct 13;353(15):1574-84. doi: 10.1056/NEJMcps050929. PMID 16221780
- [Background] Escolar ML, Poe MD, Provenzale JM, Richards KC, Allison J, Wood S, Wenger DA, Pietryga D, Wall D, Champagne M, Morse R, Krivit W, Kurtzberg J. Transplantation of umbilical-cord blood in babies with infantile Krabbe's disease. N Engl J Med. 2005 May 19;352(20):2069-81. doi: 10.1056/NEJMoa042604. PMID 15901860

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Cell Recipients | Placebo Recipients
Started | 17 | 18
Completed | 14 | 15
Not Completed | 3 | 3
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Cell Recipients | Placebo Recipients | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 18 | 35
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 16 | 17 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Survival at One Year
Description: Number of participants alive at one year.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Cell Recipients | Placebo Recipients
Number analyzed (Participants) | 17 | 18
Participants | 16 | 17

2. Primary Outcome: Number of Participants With Bayley III Scores in All Three Domains > or Equal to 85
Description: The Bayley is a standardized, norm-referenced measure that assesses development in Cognitive, Language and Motor domains. Composite standard scores can be derived that have a mean of 100 and a standard deviation of 15.
Time Frame: 1 year
Population: Participants with known one year outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Cell Recipients | Placebo Recipients
Number analyzed (Participants) | 14 | 15
Participants | 12 | 6
Statistical Analysis 1: Comparison: Intervention Cell Recipients vs Placebo Recipients; Test type: Other; p = 0.06, Fisher Exact

3. Secondary Outcome: Mortality Rate
Description: (Number of participants who died/total number of participants) x 100
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Intervention Cell Recipients | Placebo Recipients
Number analyzed (Participants) | 17 | 18
percentage of participants | 5.88 | 5.56

4. Secondary Outcome: Number of Subjects Who Experience Seizures
Time Frame: During hospitalization, approximately 4-92 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Cell Recipients | Placebo Recipients
Number analyzed (Participants) | 17 | 18
Participants | 6 | 6

5. Secondary Outcome: Number of Subjects Who Require iNO (Inhaled Nitric Oxide) Use
Time Frame: During hospitalization, approximately 4-92 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Cell Recipients | Placebo Recipients
Number analyzed (Participants) | 17 | 18
Participants | 3 | 2

6. Secondary Outcome: Number of Subjects Who Require ECMO
Description: ECMO (extracorporeal membrane oxygenation) is a technique of providing prolonged cardiac and respiratory support to persons whose heart and lungs are unable to provide an adequate amount of gas exchange or perfusion to sustain life.
Time Frame: During hospitalization, approximately 4-92 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Cell Recipients | Placebo Recipients
Number analyzed (Participants) | 17 | 18
Participants | 0 | 0

7. Secondary Outcome: Number of Subjects Who Require Gastrostomy Tube (G-tube) Feeding
Time Frame: During hospitalization, approximately 4-92 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Cell Recipients | Placebo Recipients
Number analyzed (Participants) | 17 | 18
Participants | 2 | 3

8. Secondary Outcome: Number of Subjects Who Are Discharged on Anti-epileptic Medication
Time Frame: At hospital discharge, approximately 4-92 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Cell Recipients | Placebo Recipients
Number analyzed (Participants) | 17 | 18
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention Cell Recipients | Placebo Recipients
All-Cause Mortality (participants affected / at risk) | 1/17 | 1/18
Serious Adverse Events (participants affected / at risk) | 1/17 | 2/18
Other Adverse Events (participants affected / at risk) | 1/17 | 3/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Cell Recipients (N=17) | Placebo Recipients (N=18)
Death neonatal (General disorders) | 1 | 1
Necrotizing Enterocolitis (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Cell Recipients (N=17) | Placebo Recipients (N=18)
Cord blood positive culture (Infections and infestations) | 1 | 0
Seizures (Nervous system disorders) | 0 | 2
Hypertension (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT02612155/Prot_SAP_000.pdf